CLINICAL TRIAL: NCT03947021
Title: Developing Mathematical Methods for Non-invasive Reconstruction of Electrical Heart Activity From Body-surface Electrocardiograms and a CT-based Torso-heart Geometry
Brief Title: Developing Methods for Reconstructing Electrical Heart Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: METC 11-2-043; NHS 2007T51 (Other Grant/Funding Number: Netherlands Heart Foundation)
Record Dates: First submitted 2012-11-21; First posted 2019-05-13 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Heart Diseases; Cardiac Conduction Defect
Keywords: Electrocardiography; Body Surface Potential Mapping; Computational Biology
MeSH Terms: conditions — Heart Diseases; Cardiac Conduction System Disease | interventions — Body Surface Potential Mapping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BSPM-only group (Experimental): Participants will only receive body-surface potential mapping (BSPM) with an extensive electrode set (256 electrodes).
  Interventions: Device: Body-surface potential mapping
- CT+BSPM group (Experimental): Participants will receive body-surface potential measurements (BSPM) and a CT scan. These data will allow for non-invasive reconstruction of electrical potentials at the heart surface.
  Interventions: Radiation: Computed tomography (CT) scan; Device: Body-surface potential mapping

INTERVENTIONS:
Radiation: Computed tomography (CT) scan — A CT scan of thorax and heart will be performed in the CT+BSPM group.
  Arms: CT+BSPM group
Device: Body-surface potential mapping — Measurement of 256-lead body-surface electrocardiogram

SUMMARY:
Non-invasive reconstruction of electrical heart activity can yield important scientific and clinical insights in cardiac rhythm disorders. In this study, The investigators aim at developing methods for reconstructing electrical heart activity non-invasively, and to use these methods to investigate cardiac rhythm disorders to answer clinical and scientific questions.

ELIGIBILITY:
Overall Inclusion Criteria:

* 18 years or older
* able to provide informed consent
* Conditions that might alter electrical conduction properties in the heart, including (but not limited to): Brugada syndrome (BS), Arrhythmogenic right ventricular cardiomyopathy (ARVC), demonstrated ventricular arrhythmias (resuscitation, (non)sustained ventricular tachycardia, ventricular fibrillation)
* Implanted cardiac device, such as pacemaker or implantable cardioverter defibrillator

Additional Inclusion Criteria for group 1 (CT group):

- Existing medical indication for a cardiac CT scan unrelated to this research

There are no additional inclusion criteria for group 2 (no-CT group).

Exclusion Criteria:

- Known strong reaction against electrode attachment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Epicardial potentials | Day one, direct measurement
  Primary outcome data include reconstructed electrical heart activity such as:
  - epicardial potentials (units: millivolts [mV])
  These outcome data are obtained at the moment of inclusion.
  The primary outcome measures are a comparison of the primary outcome data with invasive outcome data available from clinical records:
  - Reconstructed epicardial potentials (mV) will be compared to selected invasive epicardial potentials (mV) obtained from catheter-based recordings or pacemaker-based recordings available as clinical data
Epicardial electrograms | Day one, direct measurement
  Primary outcome data include reconstructed electrical heart activity such as:
  - epicardial electrograms (units: millivolts [mV] over milliseconds [ms])
  These outcome data are obtained at the moment of inclusion.
  The primary outcome measures are a comparison of the primary outcome data with invasive outcome data available from clinical records:
  - Reconstructed electrograms (mV) will be compared to selected invasive epicardial electrograms (mV) obtained from catheter-based recordings or pacemaker-based recordings available as clinical data
Epicardial activation and recovery sequences | Day one, direct measurement
  Primary outcome data include reconstructed electrical heart activity such as:
  - epicardial activation and recovery isochrones (units: milliseconds [ms])
  These outcome data are obtained at the moment of inclusion.
  The primary outcome measures are a comparison of the primary outcome data with invasive outcome data available from clinical records:
  - Reconstructed activation and recovery sequences (ms) will be compared to recorded catheter-based sequences from clinical data (ms).

SECONDARY OUTCOMES:
Disease-specific differences in primary outcome measures | Day one, direct measurement
  The secondary study endpoints include disease-specific differences of the primary outcome measures, which may include abnormal (low-amplitude, fractionated) electrograms and abnormal activation and recovery sequences. Depending on the primary measure, these differences will be expressed in absolute units (mV, ms) or relative differences (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands